CLINICAL TRIAL: NCT02317796
Title: A Multi-center, Double Blind, Randomized, Placebo-controlled, Parallel Group Phase IIa Study of MLR-1023 in Adult Subjects With Uncontrolled Type 2 Diabetes
Brief Title: Adult Subjects With Uncontrolled Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melior Pharmaceuticals (Other)
Collaborators: Bukwang Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BK-MD-201
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 5-(3-methylphenoxy)-2(1H)-pyrimidinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: MLR-1023
- 100 mg q.d. (Active Comparator)
  Interventions: Drug: MLR-1023
- 100 mg b.i.d. (Active Comparator)
  Interventions: Drug: MLR-1023
- 200 mg q.d. (Active Comparator)
  Interventions: Drug: MLR-1023
- 200 mg b.i.d. (Active Comparator)
  Interventions: Drug: MLR-1023

INTERVENTIONS:
Drug: MLR-1023 — Each subject will receive an oral dose of placebo or MLR-1023 once before breakfast and either placebo (placebo and q.d. dose groups) or a second dose of MLR-1023 (b.i.d. dose groups) before dinner for 4 weeks.

SUMMARY:
A Multi-center, Double Blind, Randomized, Placebo-controlled, Parallel Group Phase IIa Study of MLR-1023 in Adult Subjects With Uncontrolled Type 2 Diabetes

DETAILED DESCRIPTION:
Objectives

1. To assess the safety, tolerability and initial anti-diabetic activity of MLR-1023 in subjects with uncontrolled mild to moderate type 2 diabetes mellitus
2. To evaluate the pharmacokinetics of MLR-1023 and the major metabolite, MLR-1023-M1 following 28 days of repeat dosing

Design and Outcomes

The study is a randomized, double blind, placebo-controlled, parallel group study of MLR-1023 in adult subjects with uncontrolled type 2 diabetes mellitus who are on diet and exercise therapy.

A subset of subjects per dose group will have additional samples analyzed to measure signs of MLR-1023.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with uncontrolled T2DM who have received diet and exercise therapy for at least 3 months prior to screening, aged ≥ 18 - ≤ 75 years
2. Females must be post-menopausal, unable to conceive, or test negative for pregnancy via blood test and use barrier contraception
3. BMI ranging from ≥ 20 to ≤ 40 kg/m2
4. Fasting plasma glucose values of up to 240 mg/dL at screening, after wash-out (visit 2) and after placebo run-in (visit 3)
5. (i) naïve or (ii) currently using and discontinued metformin or (iii) no prior exposure to anti-diabetic agents other than metformin ≥ 6 months prior to screening

Exclusion Criteria:

1. History of Type 1 diabetes
2. History of more than 1 episode of severe hypoglycemia within 6 months prior to screening, or a current diagnosis of hypoglycemia unawareness.
3. Hospitalizations or Emergency room visits that would impact patient safety or data interpretation:

   1. Due to poor glucose control in the 6 months prior to screening or
   2. Any bariatric surgical procedures for weight loss.
4. Significant change of body weight (>10%) in the 3 months before screening
5. Proliferative retinopathy or maculopathy within the 6 months before screening or requiring acute treatment, or severe neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in PPG AUC0-3h in a MMTT between Days 1 and 29. | 29 Days

SECONDARY OUTCOMES:
Change in fasting plasma glucose in dose groups from Day 1 to Day 29, Day 36 | 36 Days
Change in fructosamine level from Day 1 to Day 29 | 29 Days
Change in fasting insulin from Day 1 to Day 29 | 29 Days
Change in glycated albumin from Day 1 to Day 29 | 29 Days
Change from Day 1 to Day 29 in insulin sensitivity using HOMA-R (HOMA-R = fasting plasma insulin (mU/l) * fasting plasma glucose (mmol/l) / 22.5) | 29 Days
Changes from Day 1 to Day 29 in beta-cell function using HOMA-B (HOMA-B = 20 * fast- ￼ing plasma insulin (mU/l) / [fasting plasma glucose (mmol/l) - 3.5]) | 29 Days
Change in HbA1C between Days 1 and Day 29 | 29 Days
Changes in LDL-C, HDL-C, TG between Days 1 and Day 29 | 29 Days
Change in weight between Days 1 and Day 29 | 29 Days
Differences between placebo and MLR-1023 dose groups in PPG AUC0-3h Days 1 and 29. | 29 Days

CONTACTS AND LOCATIONS:
Overall Officials: Melior Pharmaceuticals I & Bukwang Pharm. Co., Ltd., Study Director — Melior Pharmaceuticals I & Bukwang Pharm. Co., Ltd.
Locations (1):
- Melior Pharmaceuticals I & Bukwang Pharm. Co., Ltd., USA and South Korea, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Lee MK, Kim SG, Watkins E, Moon MK, Rhee SY, Frias JP, Chung CH, Lee SH, Block B, Cha BS, Park HK, Kim BJ, Greenway F. A novel non-PPARgamma insulin sensitizer: MLR-1023 clinicalproof-of-concept in type 2 diabetes mellitus. J Diabetes Complications. 2020 May;34(5):107555. doi: 10.1016/j.jdiacomp.2020.107555. Epub 2020 Feb 2. PMID 32019723